CLINICAL TRIAL: NCT04515186
Title: Efficacy and Safety of Thermotherapy in Combination With Miltefosine Compared Iltefosine Monotherapy for the Treatment of New World Cutaneous Leishmaniasis: A Phase III, Open Label, Multicenter Randomized Trial
Brief Title: Combination, Miltefosine Monotherapy for Cutaneous Leishmaniasis in New World
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DNDi-MILT-08-CL
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2024-02

CONDITIONS: Cutaneous Leishmaniases
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — Meglumine Antimoniate; miltefosine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Initial, late responders and final cure assessments done in a blinded manner by the site clinicians at D90, D105 (if required) and D180, respectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Meglumine Antimoniate (Other): Meglumine Antimoniate, 20 mg/kg/day for 20 days parenterally. This trial arm was discontinued after protocol amendment 7. However, patients assigned to this arm before protocol amendment 7 becomes effective will continue in the study and will receive complete treatment as initially planned.
  Interventions: Drug: Meglumine Antimoniate
- Miltefosine monotherapy (Active Comparator): Miltefosine monotherapy 2.5 mg/kg/day for 28 days orally
  Interventions: Drug: Miltefosine
- Thermotherapy + miltefosine (Experimental): Thermotherapy (one session, 50⁰C for 30" applications*) + miltefosine 2.5 mg/kg/day for 21 days orally.
  Interventions: Drug: Miltefosine; Device: Thermotherapy machine

INTERVENTIONS:
Drug: Meglumine Antimoniate — Vials of a 5mL solution. Each vial contains 405 mg of Sb5+ corresponding to 8.1% Sb5+ (81 mg/mL).
  Other Names: Glucantime®
  Arms: Meglumine Antimoniate
Drug: Miltefosine — 50 mg capsule
  Other Names: Impavido®
  Arms: Miltefosine monotherapy; Thermotherapy + miltefosine
Device: Thermotherapy machine — Localized Current Field radio-frequency generating device
  Other Names: ThermoMed™
  Arms: Thermotherapy + miltefosine

SUMMARY:
This study evaluates if the combination of thermotherapy (one application, 50⁰C for 30") and 3 weeks of miltefosine is safe and have a comparable cure rate with the current recommended first line treatments comprising meglumine antimoniate for 3 weeks for the treatment of uncomplicated cutaneous leishmaniasis cases in the New World.

DETAILED DESCRIPTION:
This randomized, open label, multi-centre, non-inferiority study aims to compare that the combination of thermotherapy (one application, 50⁰C for 30") and 3 weeks of miltefosine (2.5 mg/kg/day for 21 days orally) (here after referred to as combination), is non-inferior to the current recommended first line treatment miltefosine monotherapy (2.5 mg/kg/day for 28 days orally), for uncomplicated CL cases in the New World.

Originally, the study was planned to assess the non-inferiority of the combination therapy in comparison to the current recommended first line treatments, meglumine antimoniate or miltefosine monotherapy for 28 days. However, based on the revised treatment guidelines published by WHO-PAHO in 2022 in which the use of systemic antimonial received only a conditional recommendation, principally because of its well-known toxicity, and is recommended to be used only in case where there is no other option, the study protocol amendment 7 was proposed to prematurely discontinue the inclusion of additional patients in the meglumine antimoniate arm.

Primary Objective

• To determine the non-inferior efficacy of the combination in comparison to the standard first line treatment miltefosine monotherapy as measured by the percentage of patients with initial clinical cure at Day 90.

Secondary objectives

* Assess the proportion of patients who show clinical improvement at D90 (have more or equal of 75% and less than 100% re-epithelization) and achieve 100% re-epithelization at D105 (late responders).
* Assess the proportion of relapses at D180.
* Describe the proportion of patients randomized in the meglumine antimoniate arm until its discontinuation who show initial cure at D90, clinical improvement at D90 and 100% re-epithelization at D105 and relapse at D180.
* Assess the safety and tolerability profile for each regimen (percentage of treatment discontinuation, frequency and severity, causality with each study drug and seriousness of Adverse Events (AEs)).
* Assess the time to achieve 100% re-epithelialization/ flattening of ulcerated/ non ulcerated lesions by Leishmania species.

A computer-generated randomization code will be used for patient treatment allocation to one of the three arms indicated and utilizing a 1:1:1 allocation ratio.

Patients assigned to the combination treatment will start treatment at Day 1 and have a follow-up visit on 24 hours to assess safety of thermotherapy. Hereafter, these patients are required to return at Days 7, 14, 21, 45, 63, 90, 105 (late responders only) and 180 after the beginning of treatment to assess safety and efficacy.In Brazil, women of childbearing potential are required to also return on D120 and D150 to perform blood pregnancy tests. Women with irregular menstrual cycle, should return for blood pregnancy tests every two weeks until D150.

Patients assigned to the meglumine antimoniate treatment before discontinuation of this arm becomes effective arerequired to come at Days 1, 7, 14, 21, 45, 63, 90, 105 (late responders only) and 180 after the beginning of treatment to assess safety and efficacy.

Patients assigned to the miltefosine monotherapy are required to come at Days 1, 7, 14, 21, 28, 45, 63, 90, 105 (late responders only) and 180 after the beginning of treatment to assess safety and efficacy. In Brazil, women of childbearing potential are required to also return on D120 and D150 to perform blood pregnancy tests. Women with irregular menstrual cycle, should return for blood pregnancy tests every two weeks until D150.

Patients who have 100% re-epithelization at D90 are declared cured and appointed to come to their D180 assessment. If at D90 re-epithelization of the ulcer(s) is more or equal to 75% but less than 100%, patients will be defined as having clinical improvement and will be asked to return to D105 for a late responder assessment.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, aged ≥12 and ≤60 years old (upper age limit according to local regulations), and weighing ≥ 30Kg.
* Patient with a confirmed diagnosis of CL in at least one lesion by at least one of the following methods: 1) microscopic identification of amastigotes in stained lesion tissue, or 2) demonstration of Leishmania by Polymerase Chain Reaction (PCR), or 3) positive culture for promastigotes.
* Patient has a lesion that satisfies the following criteria:

  * Lesion size ≥ 0.5 cm and ≤ 4 cm (longest diameter).
  * not located on the ear, face, close to mucosal membranes, or on a location that in the opinion of the Principal Investigator (PI) is difficult to apply the TT.
  * Patient with ≤ 4 CL lesions.
  * Duration of lesion less than 4 months by patient history.
* Patient able to give written informed consent/ assent form.
* In the opinion of the investigator, the patient is capable of understanding and complying with the protocol.

Exclusion Criteria:

* Female with a positive urine or blood pregnancy test at screening or who is breast feeding or female at fertile age who does not agree to take appropriate effective contraception during treatment period and up to D180 visit. In Brazil: female at fertile age who does not agree to use two effective methods of contraception: one barrier method and one highly effective method (defined in section 8.2.4) 30 days prior to the treatment onset and up to D180 visit.
* History of clinically significant medical problems / treatment that might interact, either negatively or positively, with treatment of cutaneous leishmaniasis including any immunocompromising condition.
* Within 8 weeks (56 days) of Day 1, received treatment for the entry lesion leishmaniasis with any medication including antimonials likely, in the opinion of the PI, to modify the course of the Leishmania infection.
* Has diagnosis or suspected diagnosis of mucocutaneous leishmaniasis based on physical exam.
* Has laboratory values at screening as follows:

  * Serum creatinine: above upper normal level*.
  * Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST): 3 times above upper normal level*.

    * Normal ranges obtained from local laboratory.
* Patient who is not willing to attend the study visits or is not able to comply with follow-up visits up to 6 months.
* Known history of addiction/ alcohol abuse.
* Hypersensitivity to miltefosine or any study medication excipients.
* Patients with Sjogren-Larson Syndrome.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 184 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
The proportion of initial clinical cure in each arm. | Day 90
  Defined for ulcerated lesions as 100% re-epithelialization of the ulcer(s) on D90 as compared to D1 and for non-ulcerated lesions as flattening and/or no signs of induration of the lesion(s) on D90 as compared to D1.

SECONDARY OUTCOMES:
The number of patients who fulfil the criteria for clinical improvement at D90 and late responders at D105. | Days 90 and 105
  Clinical improvement is defined for ulcerated lesions as more than or equal to 75% but less than 100% re-epithelization of the ulcer(s) as compared to D1, and for non-ulcerated lesions as more than or equal to 75% but less than 100% of flattening and/ or signs of induration of the lesion(s) as compared to D1.
  Late responders isdefined for ulcerated lesions as 100% re-epithelialization of the ulcer(s) on D105 compared to D1, and for non-ulcerated lesions as 100% of flattening and/or no signs of induration of the lesion(s) on D105 as compared to D1.
The number of patients who fulfil the criteria of initial cure at D90 or late responders at D105 and have no relapse by D180 (final cure). | Day 180
Percentage of treatment discontinuation, frequency, severity, causality with each study drug and seriousness of AEs by treatment group. | Through study completion, i.e up to 6 months
Proportion of lesions with 100% re-epithelialization/flattening at each measurement time point by Leishmania sp. | Days 7, 14 and 21. At end of treatment (days 21 or 28), and at days 45, 63, 90, 105 and 180.
The number of patients randomized in the meglumine antimoniate arm until its discontinuation who fulfill the criteria of initial cure at D90 or late responders at D105 and have no relapse by D180 (final cure). | Day 180

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Machado, Principal Investigator — Federal University of Bahia; Marcia Hueb, Principal Investigator — Julio Muller University Hospital Federal University of Mato Grosso; Fiorela Yuly Alvarez Romero, Principal Investigator — Universidad Peruana Cayetano Heredia; Juan Miguel Pascale, Principal Investigator — Instituto Conmemorativo Gorgas de Estudios de la Salud; Jaime Soto, Principal Investigator — Fundación Nacional de Dermatología; Glaucia Cota, Principal Investigator — Instituto René Rachou Oswaldo Cruz Foundation- FIOCRUZ MINAS
Locations (6):
- Fundación Nacional de Dermatología, Santa Cruz de la Sierra, Bolivia
- Brazil (3):
  - Instituto René Rachou Oswaldo Cruz Foundation- FIOCRUZ MINAS, Belo Horizonte, Minas Gerais
  - Julio Muller University Hospital Federal University of Mato Grosso, Cuiabá
  - Federal University of Bahia Immunology Department, Salvador
- Instituto Conmemorativo Gorgas de Estudios de la Salud, Panama City, Provincia de Panamá, Panama
- Universidad Peruana Cayetano Heredia, Lima, Peru

IPD SHARING:
Plan to Share IPD: No